CLINICAL TRIAL: NCT00942825
Title: Phase II Study of a Triplet Combination of CBP501, Pemetrexed and Cisplatin as First Line Treatment in Patients With Stage IV Non-squamous Non Small Cell Lung Cancer (NSCLC)
Brief Title: Triplet Combination First Line Treatment in Non Small Cell Lung Cancer (NSCLC)
Acronym: CBP08-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CanBas Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBP08-02
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Non-squamous Non Small Cell Lung Cancer
Keywords: NSCL; non-squamous non small cell lung cancer; Lung Cancer; Lung; non-squamous; metastatic; pleural effusion; Stage IIIb; Stage IV; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Pleural Effusion | interventions — Cdc25C phosphatase (211-221); Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A CBP501 +Cisplatin + Pemetrexed (Experimental): CBP501 25 mg/m2 + Cisplatin 75 mg/m2 + Pemetrexed 500mg/m2
  Interventions: Drug: CBP501 + Cisplatin + Pemetrexed
- B Cisplatin + Pemetrexed (Active Comparator): Cisplatin + Pemetrexed
  Interventions: Drug: Cisplatin + Pemetrexed

INTERVENTIONS:
Drug: CBP501 + Cisplatin + Pemetrexed — CBP501, pemetrexed and cisplatin will be administered on the same day (Day 1), every 3 weeks for a maximum of six cycles. A cycle is considered to be 3 weeks (21 days).
  1. CBP501 25 mg/m² will be administered as an i.v. infusion of 1 hour.
  2. Pemetrexed 500 mg/m² will be administered as an i.v. infusion over 10 minutes, immediately after the CBP501 infusion.
  3. Cisplatin 75 mg/m² will be administered as a 1-hour i.v. infusion immediately after the pemetrexed infusion.
  Other Names: CBP501 + CDDP + Alimta
  Arms: A CBP501 +Cisplatin + Pemetrexed
Drug: Cisplatin + Pemetrexed — Pemetrexed and cisplatin will be administered on the same day (Day 1), every 3 weeks for a maximum of six cycles. A cycle is considered to be 3 weeks (21 days).
  1. Pemetrexed 500 mg/m² will be administered as an i.v. infusion over 10 minutes.
  2. Cisplatin 75 mg/m² will be administered as a 1-hour i.v. infusion immediately after the pemetrexed infusion.
  Other Names: CDDP + Alimta
  Arms: B Cisplatin + Pemetrexed

SUMMARY:
This is a randomized, open-label, multicenter, phase II study to compare a triplet combination of CBP501, pemetrexed and cisplatin with pemetrexed/cisplatin when administered to patients with locally advanced (stage IIIB with malignant pleural effusion or pericardial effusion) or metastatic (stage IV) non-squamous NSCLC as consecutive i.v. infusions according to a once-every-3-weeks schedule.

The protocol will evaluate full-dose cisplatin and pemetrexed with or without CBP501. Patients will be randomized in a 1:1 ratio to pemetrexed, cisplatin and CBP501 (Arm A) or pemetrexed and cisplatin (Arm B). Randomization will be stratified according to whether or not patients are eligible for bevacizumab therapy.

Preclinical and clinical findings that support this protocol are:

* CBP501 has exhibited interesting preclinical activity in various lung cancer cell lines.
* Synergism was documented with CBP501/cisplatin in the preclinical studies with lung cancer cell lines.
* The dose-limiting toxicity (DLT) of CBP501 was rapid onset allergic reaction, as was suggested by preclinical toxicology. Other toxicities were quite limited. No evidence of potentiation of either CBP501 or cisplatin toxicity was found in the combination phase I trial, and the toxicity of the combination, primarily related to cisplatin, is manageable. It is expected that CBP501 and pemetrexed will display non-overlapping toxicity profiles in combination, given that hematological toxicity and gastrointestinal toxicity are the principal toxicity types of the latter.
* Given the acceptable safety of the cisplatin/ pemetrexed combination, it is anticipated that the addition of CBP501 to this combination can be evaluated without excessive risk in the phase II programs.
* The phase I study of CBP501 in combination with pemetrexed/cisplatin (phase I part of the mesothelioma program) did not show DLTs or evidence of enhancement of toxicities with the triplet combination. The RD of CBP501 25 mg/m², cisplatin 75 mg/m² and pemetrexed 500 mg/m² is currently in use in the phase II study with first line mesothelioma patients.
* Hints of activity were observed during the phase I study with CBP501 and cisplatin.
* No pharmacokinetics (PK) interaction was documented between cisplatin and CBP501.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, phase II study to compare a triplet combination of CBP501, pemetrexed and cisplatin with pemetrexed/cisplatin when administered to patients with locally advanced (stage IIIB with malignant pleural effusion or pericardial effusion) or metastatic (stage IV) non-squamous NSCLC as consecutive i.v. infusions according to a once-every-3-weeks schedule.

The protocol will evaluate full-dose cisplatin and pemetrexed with or without CBP501. Patients will be randomized in a 1:1 ratio to pemetrexed, cisplatin and CBP501 (Arm A) or pemetrexed and cisplatin (Arm B). Randomization will be stratified according to whether or not patients are eligible for bevacizumab therapy.

The combination of cisplatin/pemetrexed has come to be recognized as the new standard of care for patients with untreated, unresectable malignant pleural mesothelioma (MPM) and untreated NSCLC non-squamous cell histology.

Preclinical and clinical findings that support this protocol are:

* CBP501 has exhibited interesting preclinical activity in various lung cancer cell lines.
* Synergism was documented with CBP501/cisplatin in the preclinical studies with lung cancer cell lines.
* The dose-limiting toxicity (DLT) of CBP501 was rapid onset allergic reaction, as was suggested by preclinical toxicology. Other toxicities were quite limited. No evidence of potentiation of either CBP501 or cisplatin toxicity was found in the combination phase I trial, and the toxicity of the combination, primarily related to cisplatin, is manageable. It is expected that CBP501 and pemetrexed will display non-overlapping toxicity profiles in combination, given that hematological toxicity and gastrointestinal toxicity are the principal toxicity types of the latter.
* Given the acceptable safety of the cisplatin/ pemetrexed combination, it is anticipated that the addition of CBP501 to this combination can be evaluated without excessive risk in the phase II programs.
* The phase I study of CBP501 in combination with pemetrexed/cisplatin (phase I part of the mesothelioma program) did not show DLTs or evidence of enhancement of toxicities with the triplet combination. The RD of CBP501 25 mg/m², cisplatin 75 mg/m² and pemetrexed 500 mg/m² is currently in use in the phase II study with first line mesothelioma patients.
* Hints of activity were observed during the phase I study with CBP501 and cisplatin.
* No pharmacokinetics (PK) interaction was documented between cisplatin and CBP501.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures
* Histologically or cytologically confirmed diagnosis of non-squamous non small cell lung cancer (NSCLC), not amenable for radical resection, stage IIIB with pleural or pericardial effusion or stage IV, who has not received previous chemotherapy or other systemic treatment
* At least one unidimensionally measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* Male or female patients aged at least 18 years
* ECOG Performance Status (PS): 0-1
* Life expectancy > 3 months
* Prior local radiotherapy is allowed if it was completed ≥ 3 weeks prior to the first dose of the study medication
* Concomitant palliative radiotherapy to an existing bone lesion for pain control is allowed
* Prior surgery is allowed if it is performed at least 4 weeks prior to the first dose of study medication and patient should be fully recovered
* Adequate organ function, including the following:
* Bone marrow: white blood cell (WBC) count >= 4 x 109/L, absolute neutrophil count (ANC) >= 1.5 x 109/L, platelet count >= 100 x 109/L, hemoglobin >= 9 g/dL
* Hepatic: Bilirubin ≤ 1.5 x the upper limit of normal (ULN), aspartate transaminases (AST/SGOT) and alanine transaminases (ALT/SGPT) ≤ 2.5 x ULN (or ≤ 5 x ULN if liver metastases are present), INR ≤ 1.5 x ULN, albumin >= 3.0 g/dL
* Renal: Serum creatinine ≤ 1.5 mg/dL or creatinine clearance >= 45 mL/min (calculated according to the Cockroft and Gault formula)
* Female patients of child-bearing potential must have a negative pregnancy test and be using at least one form of contraception as approved by the Investigator for 4 weeks prior to the study and 4 months after the last dose of study drug. For the purposes of this study, child-bearing potential is defined as: "All female patients unless they are post-menopausal for at least one year or are surgically sterile"
* Male patients must use a form of barrier contraception approved by the Investigator during the study and for 4 months after the last dose of study drug
* Ability to cooperate with the treatment and follow-up

Exclusion Criteria:

* Radiation therapy to more than 30% of the bone marrow prior to entry into the study
* Histology of pure bronchioloalveolar carcinoma or neuroendocrine features in the tumor sample
* Previous treatment with chemotherapy, new biological therapies (small molecules, antibodies), immunotherapy
* Absence of measurable lesions
* An ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the Investigator
* Any previous history of another malignancy within 5 years of study entry (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix)
* Presence of any significant central nervous system (CNS) or psychiatric disorder(s) that would hamper the patient's compliance
* Evidence of peripheral neuropathy > grade 1 according to NCI-CTCAE Version 3
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry
* Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception
* Known HIV, HBV, HCV infection
* Presence of symptomatic brain metastasis. Patients with brain metastases must:
* Have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks after completion of the definitive therapy.
* Be without neurologic dysfunction that would confound the evaluation of neurologic and other AEs
* Inability or unwillingness to take folic acid, vitamin B12 or corticosteroids
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than aspirin dose ≤ 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such piroxicam)
* Significant weight loss (>= 10% body weight during preceding 6 weeks)
* Presence of clinically significant (by physical exam) third space fluid collections, e.g., ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takumi Kawabe, MD, PhD, Study Director — CanBas Co. Ltd.
Locations (3):
- United States (3):
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - Mary Crowley Cancer Research Centers, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro GI, Tibes R, Gordon MS, Wong BY, Eder JP, Borad MJ, Mendelson DS, Vogelzang NJ, Bastos BR, Weiss GJ, Fernandez C, Sutherland W, Sato H, Pierceall WE, Weaver D, Slough S, Wasserman E, Kufe DW, Von Hoff D, Kawabe T, Sharma S. Phase I studies of CBP501, a G2 checkpoint abrogator, as monotherapy and in combination with cisplatin in patients with advanced solid tumors. Clin Cancer Res. 2011 May 15;17(10):3431-42. doi: 10.1158/1078-0432.CCR-10-2345. Epub 2011 Jan 10. PMID 21220472
- [Background] Mine N, Yamamoto S, Saito N, Yamazaki S, Suda C, Ishigaki M, Kufe DW, Von Hoff DD, Kawabe T. CBP501-calmodulin binding contributes to sensitizing tumor cells to cisplatin and bleomycin. Mol Cancer Ther. 2011 Oct;10(10):1929-38. doi: 10.1158/1535-7163.MCT-10-1139. Epub 2011 Aug 10. PMID 21831962
- [Background] Sha SK, Sato T, Kobayashi H, Ishigaki M, Yamamoto S, Sato H, Takada A, Nakajyo S, Mochizuki Y, Friedman JM, Cheng FC, Okura T, Kimura R, Kufe DW, Vonhoff DD, Kawabe T. Cell cycle phenotype-based optimization of G2-abrogating peptides yields CBP501 with a unique mechanism of action at the G2 checkpoint. Mol Cancer Ther. 2007 Jan;6(1):147-53. doi: 10.1158/1535-7163.MCT-06-0371. PMID 17237275
- [Background] Suganuma M, Kawabe T, Hori H, Funabiki T, Okamoto T. Sensitization of cancer cells to DNA damage-induced cell death by specific cell cycle G2 checkpoint abrogation. Cancer Res. 1999 Dec 1;59(23):5887-91. PMID 10606229
- [Background] Matsumoto Y, Shindo Y, Takakusagi Y, Takakusagi K, Tsukuda S, Kusayanagi T, Sato H, Kawabe T, Sugawara F, Sakaguchi K. Screening of a library of T7 phage-displayed peptides identifies alphaC helix in 14-3-3 protein as a CBP501-binding site. Bioorg Med Chem. 2011 Dec 1;19(23):7049-56. doi: 10.1016/j.bmc.2011.10.004. Epub 2011 Oct 7. PMID 22032894

RESULTS

PARTICIPANT FLOW:
Groups:
- A CBP501 +Cisplatin + Pemetrexed: CBP501 25 mg/m2 + Cisplatin 75 mg/m2 + Pemetrexed 500mg/m2
  CBP501 + Cisplatin + Pemetrexed: CBP501, pemetrexed and cisplatin will be administered on the same day (Day 1), every 3 weeks for a maximum of six cycles. A cycle is considered to be 3 weeks (21 days).
  1. CBP501 25 mg/m² will be administered as an i.v. infusion of 1 hour.
  2. Pemetrexed 500 mg/m² will be administered as an i.v. infusion over 10 minutes, immediately after the CBP501 infusion.
  3. Cisplatin 75 mg/m² will be administered as a 1-hour i.v. infusion immediately after the pemetrexed infusion.
- B Cisplatin + Pemetrexed: Cisplatin + Pemetrexed
  Cisplatin + Pemetrexed: Pemetrexed and cisplatin will be administered on the same day (Day 1), every 3 weeks for a maximum of six cycles. A cycle is considered to be 3 weeks (21 days).
  1. Pemetrexed 500 mg/m² will be administered as an i.v. infusion over 10 minutes.
  2. Cisplatin 75 mg/m² will be administered as a 1-hour i.v. infusion immediately after the pemetrexed infusion.
Period: Overall Study
Arm/Group | A CBP501 +Cisplatin + Pemetrexed | B Cisplatin + Pemetrexed
Started | 97 | 98
Completed | 97 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A CBP501 +Cisplatin + Pemetrexed | B Cisplatin + Pemetrexed | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.66) | 60.6 (9.03) | 60.6 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 36 | 87
  Male | 46 | 62 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 75 | 88 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is Progression Free Survival, Analyzed in the Treated Population. PFS is Assessed From Randomization Until Either Tumor Progression, as Per RECIST Criteria, or Until Death Due to Any Reason.
Time Frame: 15 June 2009 to 30 September 2012
Population: Treated population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A CBP501 +Cisplatin + Pemetrexed | B Cisplatin + Pemetrexed
Number analyzed (Participants) | 97 | 98
days | 140 [107 to 171] | 165 [132 to 186]

ADVERSE EVENTS:
Arm/Group | A CBP501 +Cisplatin + Pemetrexed | B Cisplatin + Pemetrexed
Serious Adverse Events (participants affected / at risk) | 37/97 | 38/98
Other Adverse Events (participants affected / at risk) | 58/97 | 53/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A CBP501 +Cisplatin + Pemetrexed (N=97) | B Cisplatin + Pemetrexed (N=98)
anemia (Blood and lymphatic system disorders) | 11 | 11
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
leukopenia (Blood and lymphatic system disorders) | 1 | 4
neutropenia (Blood and lymphatic system disorders) | 9 | 9
pancytopenia (Blood and lymphatic system disorders) | 1 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
atrial flutter (Cardiac disorders) | 0 | 1
cadiac arrest (Cardiac disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 1
GI hemorrage (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 3
peritonitis (Gastrointestinal disorders) | 1 | 0
retching (Gastrointestinal disorders) | 1 | 0
upper GI hemorrage (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 2
asthenia (General disorders) | 4 | 1
fatigue (General disorders) | 2 | 5
infusion related reaction (General disorders) | 1 | 0
infusion site reaction (General disorders) | 1 | 0
malaise (General disorders) | 1 | 0
hypersensitivity (Immune system disorders) | 1 | 0
cellulitis (Infections and infestations) | 0 | 1
infusion site cellulitis (Infections and infestations) | 1 | 0
peritonitis bacterial (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 0 | 1
ALT increased (Investigations) | 0 | 1
AST increased (Investigations) | 0 | 1
blood creatinine increased (Investigations) | 0 | 1
blood urea increased (Investigations) | 0 | 1
INR increased (Investigations) | 1 | 0
decreased apetite (Metabolism and nutrition disorders) | 3 | 4
dehydration (Metabolism and nutrition disorders) | 2 | 2
failure to thrive (Metabolism and nutrition disorders) | 1 | 0
hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
hypokalemia (Metabolism and nutrition disorders) | 1 | 3
hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 2 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
headache (Nervous system disorders) | 1 | 0
hemorrhagic stroke (Nervous system disorders) | 0 | 1
ischemic stroke (Nervous system disorders) | 0 | 1
syncope (Nervous system disorders) | 0 | 1
depressed mood (Psychiatric disorders) | 0 | 1
insomnia (Psychiatric disorders) | 1 | 0
psychotic disorder (Psychiatric disorders) | 1 | 0
renal failure acute (Renal and urinary disorders) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1
aortic thrombus (Vascular disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 1
hypertension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A CBP501 +Cisplatin + Pemetrexed (N=97) | B Cisplatin + Pemetrexed (N=98)
anemia (Blood and lymphatic system disorders) | 19 | 27
leukopenia (Blood and lymphatic system disorders) | 7 | 8
neutropenia (Blood and lymphatic system disorders) | 16 | 12
lacrimation increased (Eye disorders) | 6 | 6
constipation (Gastrointestinal disorders) | 16 | 13
diarrhea (Gastrointestinal disorders) | 9 | 8
dyspepsia (Gastrointestinal disorders) | 3 | 6
nausea (Gastrointestinal disorders) | 44 | 41
vomiting (Gastrointestinal disorders) | 24 | 25
asthenia (General disorders) | 15 | 21
chest pain (General disorders) | 7 | 8
fatigue (General disorders) | 21 | 20
infusion related reaction (General disorders) | 58 | 0
mucosal inflamation (General disorders) | 3 | 6
oedema peripheral (General disorders) | 6 | 3
pyrexia (General disorders) | 4 | 6
blood creatinine increased (Investigations) | 7 | 11
cleatinine clearance decreased (Investigations) | 6 | 1
hemoglobin decreased (Investigations) | 6 | 2
weight decreased (Investigations) | 5 | 4
decreased appetite (Metabolism and nutrition disorders) | 23 | 19
hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 5
hypomagnesemia (Metabolism and nutrition disorders) | 3 | 5
arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5
dizziness (Nervous system disorders) | 6 | 5
headache (Nervous system disorders) | 4 | 10
neuropathy peripheral (Nervous system disorders) | 9 | 4
insomnia (Psychiatric disorders) | 8 | 7
cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11
dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
alopecia (Skin and subcutaneous tissue disorders) | 4 | 8
rash (Skin and subcutaneous tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No